CLINICAL TRIAL: NCT05945459
Title: The Effect of High-calorie Density Formula Versus Standard Formula in Calorie Intake, Nutritional Status, and Clinical Outcomes Among Infants Who Underwent Congenital Heart Disease Surgery: A Randomized, Double-blind Controlled Trial
Brief Title: The Effect of High-Calorie Formula on Nutritional and Clinical Outcomes Among Infants After Congenital Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Principal Investigator, Eva M Marwali,MD, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LB.02.01/VII/214/KEP.036/2017
Record Dates: First submitted 2023-06-14; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Congenital Heart Disease in Children; Malnutrition, Child
Keywords: anthropometry; congenital heart disease; infant formula; nutritional status; randomized controlled trial
MeSH Terms: conditions — Child Nutrition Disorders; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): High-calorie density formula (1 kcal/ml)
  Interventions: Dietary Supplement: High-calorie density formula (1 kcal/ml)
- Control arm (Placebo Comparator): Standard formula (0.67 kcal/ml)
  Interventions: Dietary Supplement: Standard formula (0.67 kcal/ml)

INTERVENTIONS:
Dietary Supplement: High-calorie density formula (1 kcal/ml) — The dose is started from 20ml/kg/day divided into 8 feeds and increased by 20ml/kg/day until the feeding goal is reached (120-150ml/kg/day) during hospitalization. The intervention is then continued after discharge for 3 months (ad libitum).
  Arms: Intervention arm
Dietary Supplement: Standard formula (0.67 kcal/ml) — The dose is started from 20ml/kg/day divided into 8 feeds and increased by 20ml/kg/day until the feeding goal is reached (120-150ml/kg/day) during hospitalization. The intervention is then continued after discharge for 3 months (ad libitum).
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to compare the effect of high-calorie density formula (HDF) and standard formula (SF) in infants with congenital heart surgery. The main questions it aims to answer are:

1. Is there any difference in nutritional status between both groups after 3 months?
2. Is there any difference in calorie intake per day between both groups during hospitalization?
3. Is there any difference in clinical outcomes (mortality, duration of using mechanical ventilation, length of stay, and events of side effects) between both groups?

A group of participants will be given HDF (1 kcal/ml) from enrollment until three months. Researchers will compare them to the group of participants who are given SF (0.67 kcal/ml) to see if there is any difference in nutritional status, calorie intake, and other clinical outcomes between the two groups.

DETAILED DESCRIPTION:
The study is a randomized, double-blind controlled trial to compare the efficacy of HDF formula compared to SF in nutritional and clinical outcomes among infants who had congenital heart surgery in Harapan Kita National Cardiovascular Centre (HKNCC), Jakarta, Indonesia.

The researchers use consecutive sampling to include eligible infants and obtain informed consent from the parent or legal guardian of infants who fulfilled the eligibility criteria. Block randomization is done by a research assistant, and then the allocation is prepared using a sealed envelope to assign infants into HDF and SF groups.

Participants are then assessed by a multi-professional team and given enteral feeds based on local guidelines. Routine follow-up is done at 2 weeks, 1 month, 2 months, and 3 months after the intervention to record weight, length, and any episode of complication or adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient of less than 1 year of age who underwent congenital heart surgery procedure in Harapan Kita National Cardiovascular Center
* Risk adjustment for congenital heart surgery (RACHS) score 2-4
* Patients who do not get exclusive breastfeeding due to any cause

Exclusion Criteria:

* History of prematurity (<37 weeks gestational age)
* Formula intolerance or cow milk protein allergy
* Lethal chromosome abnormality
* Galactosemia
* Gastrointestinal malformation or obstruction
* Renal failure
* Liver disease
* Metabolic abnormalities
* Need for extracorporeal membrane oxygenation

Drop-out

* Patients who develop diarrhea for more than 5 days during the study period despite getting adequate therapy
* Patients who need prolonged total parenteral nutrition (e.g., gastrointestinal bleeding due to any cause, chylothorax, etc.)
* Patients with necrotizing enterocolitis during the study period

Ages: 14 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2019-11-03 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Nutritional status | After 3 months of intervention
  Numeric data of weight-for-length z-score (WLZ), length-for-age z-score (LAZ) and weight-for-age z-score (WAZ) based on the 2006 World Health Organization (WHO) Child Growth Standard

SECONDARY OUTCOMES:
Calorie intake | From the date of randomization to the date of discharge, assessed up to 3 months
  Numeric data of the infants' total calorie intake (kcal/kg/day) during hospitalization
Weight | After 1, 2, and 3 months of intervention
  Numeric data of absolute weight (kg)
Length | After 1, 2, and 3 months of intervention
  Numeric data of absolute length (cm)
Weight-for-age z-score changes | From the date of randomization to after 1, 2, and 3 months of intervention
  Difference of weight-for-age z-score based on The 2006 WHO Child Growth Standard
Length-for-age z-score changes | From the date of randomization to after 1, 2, and 3 months of intervention
  Difference of length-for-age z-score based on The 2006 WHO Child Growth Standard
Weight-for-length z-score changes | From the date of randomization to after 1, 2, and 3 months of intervention
  Difference of weight-for-length z-score based on The 2006 WHO Child Growth Standard
Malnutrition risk | After 1, 2, and 3 months of intervention
  Risk ratios of malnutrition, defined as weight-for-length <-2 based on 2006 WHO Child Growth Standard
Mortality | Through study completion, an average of 3 months
  The event proportion of mortality (%)
Duration of mechanical ventilation | From the date of randomization to the date of hospital discharge, assessed up to 3 months
  The difference of mechanical ventilation duration (hours)
Length of stay | From the date of randomization to the date of discharge, assessed up to 3 months
  The difference of lengths of stay in intensive care unit and hospital (days)
Side effects | From the date of randomization to the date of hospital discharge, assessed up to 3 months
  The event proportion (%) of vomiting, diarrhea, gastrointestinal bleeding, constipation, and >50% residual gastric content

CONTACTS AND LOCATIONS:
Overall Officials: Reni Fitriasari, MD, Principal Investigator — National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No